CLINICAL TRIAL: NCT05948410
Title: How Does the Mood of the Patients Change Before and After the Invasive Urodynamic Study?
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Koç University (Other)
Responsible Party: Principal Investigator, Ersin Köseoglu, MD, Koç University
Other Study IDs: KocUrol3
Record Dates: First submitted 2023-07-09; First posted 2023-07-17 (Actual); Last update posted 2023-07-17 (Actual); Status verified 2023-07

CONDITIONS: Lower Urinary Tract Symptoms; Mood Change; Diagnosis
Keywords: invasive urodynamic study; mood
MeSH Terms: conditions — Lower Urinary Tract Symptoms; Disease | interventions — Perceived Stress Scale

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Week
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Study Group: Patients with an indication of invasive urodynamic study
  Interventions: Behavioral: The State-Trait Anxiety Inventory (STAI); Behavioral: Perceived Stress Scale; Behavioral: Visual Analog Scale

INTERVENTIONS:
Behavioral: The State-Trait Anxiety Inventory (STAI) — The State-Trait Anxiety Inventory (STAI) is a psychological inventory consisting of 40 self-report items on a 4-point Likert scale. The STAI measures two types of anxiety - state anxiety and trait anxiety. Higher scores are positively correlated with higher levels of anxiety.
Behavioral: Perceived Stress Scale — The Perceived Stress Scale (PSS) is the most widely used psychological instrument for measuring the perception of stress. It is a measure of the degree to which situations in one's life are appraised as stressful. Items were designed to tap how unpredictable, uncontrollable, and overloaded respondents find their lives. The scale also includes a number of direct queries about current levels of experienced stress. PSS scores are obtained by reversing responses (e.g., 0 = 4, 1 = 3, 2 = 2, 3 = 1 & 4 = 0) to the four positively stated items (items 4, 5, 7, & 8) and then summing across all scale items. A short 4 item scale can be made from questions 2, 4, 5 and 10 of the PSS 10 item scale
Behavioral: Visual Analog Scale — The visual analogue scale (VAS) is a psychometric response scale that can be used in questionnaires. It is a measurement instrument for subjective characteristics or attitudes that cannot be directly measured. When responding to a VAS item, respondents specify their level of agreement to a statement by indicating a position along a continuous line between two end points.

SUMMARY:
The goal of this study is to learn about the patient's perspective regarding to psychological mood before and after an invasive urodynamic study.

DETAILED DESCRIPTION:
The participants have already had an indication of an invasive urodynamic study. All patients will be given STAI, perceived stress scale and VAS forms just before, after and 1-week following an invasive urodynamic study. The scores will be compared.

ELIGIBILITY:
Inclusion Criteria:

* Patients with an invasive urodynamic study indication

Exclusion Criteria:

* Non-Turkish speakers
* Poor conscious state

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with an indication of invasive urodynamic study
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2023-10-01 (Estimated); Primary Completion 2024-10-01 (Estimated); Study Completion 2025-01-01 (Estimated)

PRIMARY OUTCOMES:
The State-Trait Anxiety Inventory (STAI) | 1 week
  Questionnaire
Visual Analogue Scale | 1 week
  Questionnaire
Perceived Stress Scale | 1 week
  Questionnaire

IPD SHARING:
Plan to Share IPD: No